CLINICAL TRIAL: NCT05303142
Title: Comparison of Novel Putative Risk Factors for Exertional Heat Illness Between a Military Patient Cohort and Matched Control Cohort During Exercise Heat Stress
Brief Title: Comparing Exertional Heat Illness Risk Factors Between Patients and Controls
Status: Completed | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Liverpool John Moores University (Other); Institute of Naval Medicine (UK) (Unknown); Headquarters Army Recruiting and Initial Training Command (UK) (Unknown); Public Health Wales (Other Government)
Responsible Party: Principal Investigator, Jo Corbett, Principal Investigator, University of Portsmouth
Other Study IDs: 209321
Record Dates: First submitted 2022-02-03; First posted 2022-03-31 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Exertional Heat Illness
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva; plasma; stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with a history of EHI: Service personnel who have a history of EHI.
  Interventions: Other: Heat Tolerance Assessment
- Control participants without a history of EHI: Matched control participants with no history of EHI. They will be matched to the experimental group for parameters that are known to influence thermoregulatory responses to exercise heat-stress.
  1. Relative aerobic fitness (V̇O2max; ml∙kg-1∙min-1)
  2. Body mass (kg)
  3. Body surface area (m2)
  4. Age
  5. Sex
  Interventions: Other: Heat Tolerance Assessment

INTERVENTIONS:
Other: Heat Tolerance Assessment — 60-90 minutes exercise in hot (34 °C; 45% R.H.) conditions at 60%VO2max

SUMMARY:
The arduous nature of military training and operations require personnel to encounter high heat load, e.g., during intense physical exertion, particularly in the heat. These conditions reduce operational effectiveness and expose personnel to a risk of incapacitation and death from exertional heat illness (EHI). The primary aim of this study is to compare putative 'chronic' EHI risk factors between a cohort who have suffered a history of EHI and a control cohort with no EHI history. The secondary aim is to examine the influence of these EHI risk factors on thermoregulation during a standard heat tolerance assessment.

DETAILED DESCRIPTION:
Military training and operations present a risk of incapacitation and death from Exertional Heat Illness (EHI). However, widely accepted EHI risk factors are absent in almost half of all United Kingdom (UK) military EHI cases, indicating that a significant number of EHI cases in military personnel involve alternative risk factors. Risk factors for EHI can been classified along a spectrum ranging from acute (e.g. recent poor sleep) to chronic (e.g. low fitness), with the role of chronic risk factors supported by the observation that individuals who have suffered an EHI are at a substantially increased risk of subsequent EHI. The primary aim of this study is to compare putative 'chronic' EHI risk factors (e.g. composition of gastrointestinal (GI) microbiome, infection and inflammation, trait-like psychological factors) between a cohort who have suffered a history of EHI and a control cohort with no EHI history. The secondary aim is to examine the influence of these EHI risk factors on thermoregulation during a standard heat tolerance assessment.

ELIGIBILITY:
Inclusion Criteria:

Individuals with a history of EHI:

* Previous EHI episode
* Normal resting ECG
* Male or female
* 18 - 40 years

Control participants:

* No previous history of EHI
* Normal resting ECG
* Male or female
* 18 - 40 years

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who have experienced a recent exertional heat illness and matched controls with no previous history of exertional heat illness
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Core temperature | At 60 minutes (or test termination if earlier) of Heat Tolerance Assessment
  Measured using a rectal thermistor.
Core temperature | Rate of rise from 30 to 60 minutes (or test termination if earlier) of Heat Tolerance Assessment
  Measured using a rectal thermistor.
Diversity of gastrointestinal microbiota | Baseline
  Measured in stool sample. Assessed by alpha diversity score.
Diversity of gastrointestinal microbiota | Baseline
  Measured in stool sample. Assessed by beta diversity score.
Abundance of gastrointestinal microbiota | Baseline
  Measured in stool sample. Assessed at level of phylum.
Detection of sexually transmitted pathogens | Baseline
  Assessed from urine sample. Measured using cobas CT/NG assays.
Detection of respiratory pathogens | Baseline
  Assessed from throat swab. Measured using Allplex assays.
Detection of gastrointestinal pathogens | Baseline
  Assessed from stool swab. Measured using Allplex.
Circulating Interleukin 6 | Baseline
  Measured using ELISA
Circulating Interleukin 6 | Post Heat Tolerance Assessment (within 15 minutes of test end)
  Measured using ELISA
Circulating C-Reactive Protein | Baseline
  Measured using ELISA
Circulating C-Reactive Protein | Post Heat Tolerance Assessment (within 15 minutes of test end)
  Measured using ELISA
Circulating Claudin 3 | Baseline
  Measured using ELISA
Circulating Claudin 3 | Post Heat Tolerance Assessment (within 15 minutes of test end)
  Measured using ELISA
Circulating Zonulin | Baseline
  Measured using ELISA
Circulating lipopolysaccharide binding protein | Baseline
  Measured using ELISA
Circulating lipopolysaccharide binding protein | Post Heat Tolerance Assessment (within 15 minutes of test end)
  Measured using ELISA
Circulating intestinal fatty acid binding protein | Baseline
  Measured using ELISA
Circulating intestinal fatty acid binding protein | Post Heat Tolerance Assessment (within 15 minutes of test end)
  Measured using ELISA
Gastrointestinal illness symptomology questionnaire | Baseline
  Visual analogue scale (0-10). Higher scores indicate worse symptomology
Gastrointestinal illness symptomology questionnaire | Pre Heat Tolerance Assessment
  Visual analogue scale (0-10). Higher scores indicate worse symptomology
Gastrointestinal illness symptomology questionnaire | Immediately post Heat Tolerance Assessment
  Visual analogue scale (0-10). Higher scores indicate worse symptomology
Respiratory illness symptomology, measured by Jackson common cold questionnaire | Baseline
  Higher scores indicate worse symptomology
Sleep quality and quantity, measured by Pittsburgh Sleep Quality Index | Baseline -3 days
  Higher scores indicate worse sleep
Motivation, measured by Motivation scale | Baseline -3 days
State-trait anxiety, measured by state-trait anxiety inventory form Y-2 | Baseline -3 days
Risk taking, measured by the risk-taking inventory | Baseline -3 days
Resilience, measured by the Connor-Davidson resilience scale | Baseline -3 days
Stress, measured by perceived stress scale | Baseline -3 days
Mental readiness | Baseline
  Visual analogue scale (0-100). Higher scores indicate a lower state of mental readiness.
Stress | Baseline
  Visual analogue scale (0-100). Higher scores indicate a greater state of stress.

SECONDARY OUTCOMES:
Heat rate | At 5 minute intervals during the Heat Tolerance Assessment
Thermal comfort | At 15 minute intervals during Heat Tolerance Assessment
  Modified 9 point Gagge scale. Higher scores indicate worse comfort.
Thermal sensation | At 15 minute intervals during Heat Tolerance Assessment
  Modified 9 point Gagge scale. Higher scores indicate hotter sensation
Rating of Perceived Exertion | At 15 minute intervals during Heat Tolerance Assessment
  6-20 Borg scale. Higher scores indicate higher perceived exertion
Skin Temperature | During Heat Tolerance Assessment
  Weighted mean skin temperature
Sweat rate | During Heat Tolerance Assessment
  Determined from change in nude body mass during the heat tolerance assessment

OTHER OUTCOMES:
Body mass | Baseline
Relative maximal aerobic fitness | Baseline
  Highest value measured in ml.kg-1.min-1 during a treadmill graded exercise test.
Urine osmolality | Baseline
  Measured using freezing point depression

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No